CLINICAL TRIAL: NCT02701959
Title: Growth of Lettuce With Different Content of Inorganic Nitrate as a Feeding Strategy for Placebo-controlled Nutritional Interventions to Test the Effects of Inorganic Nitrate on Human Health
Brief Title: Effect of Lettuce With Different Nitrate Contents on Blood Pressure
Acronym: LBP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15-QAD-15
Record Dates: First submitted 2016-02-17; First posted 2016-03-08 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Dietary Modification; Blood Pressure
Keywords: Nitric oxide; Dietary intervention trail

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low nitrate lettuce (Placebo Comparator): 50g of low nitrate lettuce (placebo) on single occasions
  Interventions: Dietary Supplement: Low Nitrate Lettuce
- High nitrate lettuce (Active Comparator): 50g of high nitrate lettuce (intervention) on single occasions
  Interventions: Dietary Supplement: High Nitrate Lettuce

INTERVENTIONS:
Dietary Supplement: High Nitrate Lettuce — The lettuce has been grown with high concentration of nitrogen fertilizer (150ppm) to produce the high of nitrate content in the lettuce, the nitrate content of 50 grams of high nitrate lettuce was (~530 mg nitrate derived).
  Arms: High nitrate lettuce
Dietary Supplement: Low Nitrate Lettuce — The lettuce has been grown with low concentration of nitrogen fertilizer (25ppm) to produce the low amount of nitrate in the lettuce, the nitrate content of 50 grams of high nitrate lettuce was (~3 mg nitrate derived).
  Arms: Low nitrate lettuce

SUMMARY:
Leafy vegetables are a natural source of dietary nitrate, which may reduce systolic blood pressure (BP). However, the evidence has been obtained from studies using nitrate solutions (i.e., potassium or sodium nitrate) or beetroot juice supplementation which have a suitable placebo for the design of double-blind clinical trials. However, the design of food-based nutritional interventions is complicated by the fact that an appropriate placebo treatment is not available and, therefore, it is not possible to meet the criteria for proper double-blind randomised placebo-controlled intervention trials. In addition, the biological effects of processed products such as beetroot juice or solutions with a pharmacological grade may be different from that of fresh vegetables, e.g. due to conversion of nitrate to nitrite in the mouth during chewing.

Objectives: to investigate whether two sets of lettuce specifically grown with different nitrate content but otherwise similar composition show different effects on nitrate uptake and bioavailability in humans. Additionally, the investigators also aim to design human intervention studies to investigate the effect of intake of lettuce with different nitrate content on vascular health.

These objectives will be tested by growing lettuce with different fertiliser compositions resulting in high and low nitrate content and then investigating the bioavailability and short-term effect on BP in healthy young volunteers in a double-blind cross-over design. Eligible subjects will consume one meal each of either low or high nitrate lettuce. Urine, blood and saliva samples will be collected at baseline, for 6 hours after the ingestion and then again after 24hr. Blood Pressure BP will be measured continuously for 24 hours starting at baseline. The volunteers will repeat the intervention with the second treatment.

DETAILED DESCRIPTION:
Study Design and Subjects: This study is designed as a double-blind, randomized, crossover, intervention trial in which thirty healthy young volunteers (BMI: 20-25 kg/m2), non-smoking subjects (age: 18-35 years) will be recruited. In each of two intervention periods, subjects will be asked to eat 50g of either high nitrate lettuce or low nitrate lettuce (placebo) on a single occasion (the second visit) with dietary restriction for 3 days prior to the second visit and in the 24 hr period following after the consumption, concluded with a third visit, with at least 3 weeks washout period before the second 2-day intervention period. Urine, saliva and blood samples will be collected during a 6-hour period during the second visit. Urine samples will be collected during 24h from consumption until the third visit, to assess the pharmacokinetics and bioavailability and compliance to the interventions (details in the diagram of human trial).

The primary outcomes are 24-hour BP and nitrate content in urine, plasma and saliva. Samples will be collected into tubes and then analysed in the laboratory for the nitrate content (NO3-) by gas chromatography-mass spectroscopy (GCMS). Participants will follow specific dietary and lifestyle instructions to minimise confounding effects.

Participant will receive a small honorarium after the study and reasonable travel expenses will be reimbursed.

Dietary Interventions: Participants will be asked to arrive fasting in the morning of the second (main) visit and will consume a standard meal (Chicken Hotpot from ASDA) with the same drink water at the evening before and the evening after the visit, as well as following a diet that excludes a list of specific foods containing high nitrate (rocket, spinach, other leafy vegetables, radish and beet root), cured meat, cured seafood and cured fish, mature cheese for 24hr prior to the study and fasting on the morning of the study.

Anthropometry: This includes the measurements of body weight, height and waist circumference according to standardised protocols. Procedures are safe, not invasive and induce minimal discomfort for the participants.

Body Composition: This includes the measurement of body fat and muscle using a non-invasive technique called bio impedance analysis using a leg-to-leg bioelectrical impedance device (TANITA 300 MA). The procedure is safe, non-invasive and induces minimal discomfort for the participant. The duration of the measurement is of approximately 3-5 minutes.

24-hr BP monitoring: participants will be fitted with an automated portable device to measure BP over a 24-hr period. Participants will be instructed on how to safely operate the device. The measurement are safe and minimally invasive. BP readings will be recorded every 30 minutes during day time and every hour during the night to minimise the potential impact on sleep quality.

Urine samples: The first morning void (FMV) will be collected at home (pre supplementation) and after arrival full urine samples (all that the volunteer is able to produce) at set times before and after the supplementation (between baseline and 6hr) at NU-Food research facility. Subsequent collections afterwards (between 6-12hr and 12-24 hr) will take place at home in appropriate plastic containers and the samples will be collected at the final visit 24hr after the consumption. After measuring the volume of each sample, sub samples will be stored for analysis and for calculation of pharmacokinetics.

Saliva samples: a small saliva sample (~2ml) will be collected in disposable plastic containers at baseline and at every hour for 6 hours at NU-Food research facility; and then after 9 and 12 hour at home, with the final sample taken after 24 hr.

Blood Samples: Venous blood samples (LH 6 ml) will be collected at baseline, three and six hours post supplementation of treatments and then again after 24 hr.

ELIGIBILITY:
Inclusion criteria:

The investigators aim to recruit 20 healthy young volunteers, non-smoking, male and female aged 18-35 years with a body mass index (BMI) in the range of 20 to 25 kg/m2.

Exclusion criteria (reason for exclusion):

* Current participation in other clinical investigations.
* Mouthwash users.
* Vegetarianism (likely to have very high nitrate intake)
* Dislike to lettuce consumption or inability to comply with the study diet (lack of compliance)
* Use of antihypertensive or cholesterol lowering medication.
* History of any major illness such as cancer; or cholesterol lowering medication; history of cardiovascular or peripheral vascular disease;
* History of any major illness such as cancer; a psychiatric illness; recent history of asthma, renal, liver or gastrointestinal disease.
* Use of antibiotics within previous 2 months; current or recent (within previous 6 months) significant weight loss or gain (>6% of body weight); --woman who were pregnant, lactating or wishing to become pregnant during the study.
* Previous diagnosis of type 1 or type-2 diabetes treated with insulin (modification of regulation of intermediate metabolism).
* Major surgical operations interfering with the study outcomes (systemic effects on study outcomes).
* Alcohol intake >21 units/week for men and >14 units/week women
* Non English speakers or volunteers requiring translators or interpreters (since these services are not available for this study).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour Ambulatory Blood Pressure (AMBP) | Baseline and 24 hours
  Change in Systolic and Diastolic Blood Pressure at baseline and every 30 minutes at day time and every hour at night time for 24 hours.

SECONDARY OUTCOMES:
Change in bio-availability of nitrate and nitrite in plasma | 24 hours
  Change in plasma nitrate and nitrite at baseline, 3 hours, 6 hours and 24 hours from intervention.
Change in Cyclic Guanosine Monophosphate (cGMP) in plasma samples | 24 hours
  Change in Cyclic Guanosine Monophosphate (cGMP) in plasma samples at baseline, 3 hours, 6 hours and 24 hours from intervention.
Change in bio-availability of nitrate and nitrite in urine samples | 24 hours
  Change in urinary nitrate and nitrite at baseline, 0-3, 3-6, 6-12 and 12-24 hours from intervention.
Change in bio-availability of nitrate and nitrite in saliva samples | 24 hours
  Change in salivary nitrate and nitrite at baseline, 0, 1, 2, 3, 4, 5, 6, 9, 12 and 24 hours from intervention.
Change in Antioxidant capacity of Ferric Reducing Antioxidant Power (FRAP) and Trolox Equivalent Antioxidant Capacity (TEAC) in plasma samples. | 24 hours
  Change in Antioxidant capacity of Ferric Reducing Antioxidant Power (FRAP) and Trolox Equivalent Antioxidant Capacity (TEAC) in plasma samples at baseline, 3 hours, 6 hours and 24 hours from intervention.

CONTACTS AND LOCATIONS:
Overall Officials: AFRD School, Study Director — School of Agriculture, Food and Rural development
Locations (1):
- School of Agriculture, Food and Rural Development, Newcastle upon Tyne, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
I can't share the individual participants data because of the privacy of volunteers have been participated in this study and this already been mentioned in the application form of ethical approval.

REFERENCES:
- [Derived] Qadir OK, Seal CJ, Ashor AW, Tassotti M, Mena P, Del Rio D, Siervo M, Brandt K. Double-blind controlled dietary cross-over intervention with differentially fertilised intact lettuce leaves shows acute reduction in blood pressure in young adults, associated with faster uptake of nitrate than of phenolics. Eur J Nutr. 2022 Dec;61(8):4191-4203. doi: 10.1007/s00394-022-02961-5. Epub 2022 Jul 23. PMID 35871120